CLINICAL TRIAL: NCT05468983
Title: BioHPP Hybrid Prosthesis Versus BioHPP Bar Implant Supported and Retained Overdenture Rehabilitating Edentulous Mandible
Acronym: BioHPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 686
Record Dates: First submitted 2022-03-30; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Marginal Bone Loss; Patient Satisfaction
Keywords: BioHpp; hybrid prosthesis; overdenture; bone loss
MeSH Terms: conditions — Patient Satisfaction; Bone Diseases, Metabolic | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: to compare BioHPP used as a skeletal substructure for hybrid (implant fixed, detachable) prostheses versus BioHPP bar supporting and retaining by using radiographic tracing to the marginal bone height changes around the implants, patient satisfaction can be improved.
Who Masked: Investigator
Masking Description: All the Selected patients were rehabilitated with the upper and the lower complete denture then was divided by computer randomization "using random allocation software: into two equal groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BioHpp hybrid prosthesis( fixed ) (Other): 4 implants were placed in the mandibular arch by a surgical guide, after 3 months the final prosthesis was constructed by using a digital workflow( CAD-CAM )
  Interventions: Procedure: surgical ( implants placement)
- BioHpp bar supported and retained overdenture (Other): 4 implants were placed in the mandibular arch by a surgical guide, after 3 months the final prosthesis was constructed by using a digital workflow( CAD-CAM )
  Interventions: Procedure: surgical ( implants placement)

INTERVENTIONS:
Procedure: surgical ( implants placement) — 4 implants were placed interforamen of the mandibular arch by using the surgical guide
  Other Names: Final prosthesis was constructed on the 4 implants

SUMMARY:
The biggest challenge of oral rehabilitation is the replacement of lost structures and the restoration of their function and esthetics, focusing on matching a healthy tooth.

Traditional complete dentures, implant (retained, supported) overdentures, and complete implant-supported fixed prostheses are all alternatives to the rehabilitation of the mandibular arch.

The aim of this study was to compare BioHPP used as a skeletal substructure for hybrid (implant fixed, detachable) prostheses versus BioHPP bar supporting and retaining by using radiographic tracing to the marginal bone height changes around the implants, patient satisfaction can be improved.

DETAILED DESCRIPTION:
Fourteen completely edentulous male patients were selected from the out-patient clinic, Prosthodontic Department, Faculty of Dentistry, Ain Shams University, according to certain criteria, and they were randomly allocated into two equal groups: group I: the seven patients were rehabilitated by the BioHpp hybrid prosthesis supported on four inter-foraminal implants; group II: While in group II, seven patients were rehabilitated by the BioHpp bar supported and retained overdenture.

The upper and lower complete dentures were constructed following conventional methods, and the surgical guide was constructed according to dual-scan CBCT.

the four parallel inter-foraminal implants were inserted in the mandible for each patient through used the surgical guide ( flapless technique ) After three months from the first surgery, the final prosthesis was constructed.

For Group I; BioHpp fixed hybrid prosthesis, for Group II; BioHpp bar implant-supported and retained complete overdentures were created using digital workflow CAD/CAM.

The crestal bone height loss was evaluated after six, twelve, and eighteen months from implant loading by using digital preapical radiography. Also, the patient's subjective evaluations by using a questionnaire based on the visual analog scale including five points (low dissatisfied, dissatisfied, fair, satisfied, highly satisfied) were evaluated for speech, chewing, comfort aesthetic, oral hygiene, and general satisfaction.

A comparison between groups I and II was performed by using the Chi-square test, which revealed in the results that group II was significantly lower than group I at all intervals in the mesial and distal surfaces of anterior and posterior implants. Also, the results of the patient satisfaction revealed that, after 6 months, there was an insignificant difference between them as P > 0.05 in all except oral hygiene, as satisfaction was significantly higher in group II than in group I. While, after 12 months, there was an insignificant difference between them all (P > 0.05).

ELIGIBILITY:
Inclusion Criteria:

1- sufficient inter arch distance. 2. good oral hygiene. 3. Enough bone volume in interforaminal region.

Exclusion Criteria:

1. TMJ disorders.
2. Radiotherapy or chemotherapy.
3. Diabetes mellitus
4. Uncooperative patients

Ages: 55 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All selected patients were healthy to minimize gender difference and to avoid the sex-related hormonal changes that accompany the menopausal and post-menopausal periods in females, which might affect the rate of alveolar ridge resorption
Enrollment: 14 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
bone height change around implants | from insertion ( base line) to 6 months ) , from 6 months to 12 months ,from 12 months to 18 months , from insertion to 12 months, from insertion to 18 months
  The bone loss measurements were taken using a digital preapical radiograph as follows: Two horizontal lines were drawn at the alveolar bone crest and the implant apex; the software then automatically displays the measurements in millimeters between the two lines on the screen. Subtraction was used to compute the difference in bone height. The mean of the mesial and distal readings was calculated. The software then displays the measurements in millimeters between the two lines on the screen. At each follow-up visit, the values of linear measurements were recorded in the patient's chart, and the mean value of bone height change was calculated using this data.

SECONDARY OUTCOMES:
patient satisfactions | 6 months and 18 months
  Patient satisfaction was evaluated using a questionnaire based on the visual analog scale (VAS). Patients were asked to mark their answers (amount of satisfaction). The questionnaire was given to the patients in Arabic.Six factors were rated on a 1 to 5 scale (highly satisfied = 5; satisfied = 4; fair = 3; dissatisfied = 2; highly dissatisfied = 1). The sum of the five sub-scores was then calculated, ranging from 5 to 30 (best score = 30, worst score = 5). The low range of scores indicated low satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud H El Afandy, prof, Study Director — faculty of dentistry ,Ain Shames University; Magda H Mohamed, lectu, Principal Investigator — faculty of dentistry ,Ain Shames University
Locations (1):
- Prosthodontics Department Faculty of Dentistry, Cairo, Ain Shames University, Egypt